CLINICAL TRIAL: NCT04260204
Title: Effect of Retrograde Autologous Blood Priming of Cardiopulmonary Bypass on Hemodynamic Parameters and Pulmonary Mechanics in Pediatric Cardiac Surgery
Brief Title: Effect of Retrograde Autologous Blood Priming on Pulmonary Mechanics in Pediatric Cardiac Surgery
Acronym: RAPCPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr. Hamdy Singab, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACTS004367
Record Dates: First submitted 2020-02-01; First posted 2020-02-07 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Congenital Heart Disease
Keywords: retrograde autologous priming pulmonary mechanics
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Patients were included in the study if they had left to right shunt due to volume or pressure overload
Who Masked: Participant, Investigator
Masking Description: double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde priming (Active Comparator): retrograde autologous Blood Priming of Cardiopulmonary Bypass (RAP) in young children subjected to cardiac surgery for congenital heart defects with left to right shunt associated with volume or pressure overload.
  Interventions: Procedure: Pediatric cardiac surgery
- conventional priming (Active Comparator): conventional cardiopulmonary priming in young children subjected to cardiac surgery for congenital heart defects with left to right shunt associated with volume or pressure overload.
  Interventions: Procedure: Pediatric cardiac surgery

INTERVENTIONS:
Procedure: Pediatric cardiac surgery

SUMMARY:
The present study hypothesized that beyond its hemodynamic affects,retrograde autologus blood priming of cardiopulmonary bypass (RAP) has a positive impact on hemodynamics and pulmonary mechanics subjected to cardiac surgery.

DETAILED DESCRIPTION:
This prospective randomized study analyzed the clinical records of 124 children subjected to cardiac surgery for congenital heart diseases with left to right shunt. They comprised 64 patients with RAP and 60 patients conventional cardiopulmonary bypass priming. The preoperative, intraoperative and postoperative data of the studied patients were reported.

ELIGIBILITY:
Inclusion Criteria:

* children complained of congenital heart disease with left to right shunt pressure or volume load

Exclusion Criteria:

* cyanotic heart disease

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Comparison of postoperative peak air way pressure between the studied groups | 1 hour after surgery
  peak air way pressure (Paw) in cmH2O
Comparison of postoperative air way resistance between the studied groups | 1 hour after surgery
  air way resistance (Raw) in cmH2O/L/sec.
Comparison of postoperative Plateau pressure between the studied groups | 1 hour after surgery
  Plateau pressure in cm H2O
Comparison of postoperative Lung compliance between the studied groups | 1 hour after surgery
  Lung compliance in L/cm H2O
Comparison of postoperative Tidal volume between the studied groups | 1 hour after surgery
  Tidal volume in ml

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Singab, PhD, Principal Investigator — Ain shams university faculty of medicine

IPD SHARING:
Plan to Share IPD: Yes
Pulmonary mechanics improvement in pediatric patients undergoing cardiac surgery with retrograde autologous priming
Supporting Information: CSR
Time Frame: 6 months
Access Criteria: Pediatric cardiac surgeon